CLINICAL TRIAL: NCT01957228
Title: Causative Diagnosis on Prosthetic Joint Infections: Establishment of a Comprehensive Diagnostic Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-A00960-45; 2013-28 (Other: AP HM)
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Prosthetic Joint Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bone biopsies (Experimental)
  Interventions: Procedure: bone biopsies

INTERVENTIONS:
Procedure: bone biopsies

SUMMARY:
On joint orthopaedic hardware infections are one of the most frequently encountered complications in orthopaedic surgery. However 6% of the cultures remain sterile, etiological diagnosis cannot be established despite obvious signs of infection. As part of this research project, we have developed a new strategy diagnosis including directly the use of PCR to reduce the number of negative results. This should have a major therapeutic impact in terms of timeliness and specificity of antibiotic.

Primary:

Evaluate the effectiveness of the new diagnostic strategy on etiological identification of prosthesis infections.

Hypothesis:

Minimum 6 percent increase in the number of patients with an etiological diagnosis of infection on prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is more than 18 years old.
* Patient with a prescription of a microbiologic diagnostic of Prosthetic joint infection
* Patient who do not declined to have his medical records reviewed for research
* Patient with health insurance

Exclusion Criteria:

* Patient minor (<18 years).
* Pregnant or lactating woman.
* Major under guardianship Patient.
* Patient deprived of liberty or under court order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 980 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Bone biopsies multisite | 4 years
  Increase of at least 6% of patients with an etiologic diagnosis of prosthesis infection established.

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France